CLINICAL TRIAL: NCT02097680
Title: Influence of the Aromatase Inhibitor Letrozole on Heart and Liver Function in Obese Men
Brief Title: Influence of Aromatase Inhibition on Hepatic- and Cardiac Function in Severe Obese Men
Acronym: HEPAROB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: EC/2013/912; 2013-002964-22 (EudraCT Number)
Record Dates: First submitted 2014-03-17; First posted 2014-03-27 (Estimated); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Obesity
Keywords: with disturbed glucose metabolism; without disturbed glucose metabolism
MeSH Terms: conditions — Obesity | interventions — Letrozole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Letrozole (Experimental)
  Interventions: Drug: Letrozole
- Placebo comparator (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Letrozole — One Letrozole 2.5 mg capsule every two days during four months
  Other Names: Femara
  Arms: Letrozole
Drug: Placebo — One placebo capsule every two days during four months
  Arms: Placebo comparator

SUMMARY:
It seems plausible that increased aromatase activity in obese men, as a result of a larger fat mass, is responsible for decreased levels of testosterone. Therefore aromatase inhibition increases testosterone levels, which may affect hepatic and cardiac function.

In this intervention study two groups of hypogonadal obese men are compared. Group A is treated with Letrozole 2.5 mg (aromatase inhibitor) once every two days during four months; a group with normal testosterone and low oestrogen concentrations. Group B is treated with placebo once every two days during four months; this group will retain low testosterone - and high oestrogenic concentrations.

The primary objective of the study is to evaluate effects of changed sex steroids in obese men on hepatic and cardiac function.

ELIGIBILITY:
Inclusion Criteria:

* Obese male subjects
* Planned for gastric bypass (BMI > 30 kg/m²)
* low testosterone levels
* age between 20 and 65

Exclusion Criteria:

* Primary hypogonadism or secondary hypogonadism due to genetic causes (Kallman syndrome etc.), tumours, infiltrative diseases, infections, pituitary apoplexy, trauma, critical illness, chronic systemic illness or intentional.
* Treatment with corticoids, opiates (on a daily basis), androgen- or estrogen analogs or CYP2A6 substrates (Dexmedetomidine, Ifosfamide, Methoxsalen, Miconazole, Tranylcypromine).
* Impaired renal function defined as serum-creatine > 1.5 mg/dL
* Clinically significant active cardiovascular disease including history of myocardial infarction within the past 6 months and/or heart failure (NYHA class III or IV) at the discretion of the investigator
* Cancer or any clinically significant disease or disorder, which in the investigator's opinion could interfere with the results of the trial
* Palpable prostate nodule or induration, Prostate-specific antigen (PSA) > 3 ng/mL, prostatism, untreated sleep apnea syndrome, erythrocytosis (hematocrit > 50%) or hyperviscosity. (cfr. Endocrine Society Clinical Practice Guideline by Bhasin S et al.)
* Known or suspected abuse of alcohol or narcotics

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-12; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
cardiac function parameters | after 4 months intervention
  heart function will be measured by echocardiography.
Hepatic function parameters | before intervention
  Baseline sex steroids will be measured by Liquid chromatography-mass spectrometry (LC-MS/MS) in fasting blood samples, before 10:00 am. Liver function will be analysed by a Nuclear Magnetic Resonance (NMR) recording
Hepatic function parameters | after 4 months intervention
  Baseline sex steroids will be measured by Liquid chromatography-mass spectrometry (LC-MS/MS) in fasting blood samples, before 10:00 am. Liver function will be analysed by a Nuclear Magnetic Resonance (NMR) recording
cardiac function parameters | before intervention
  heart function will be measured by echocardiography.

SECONDARY OUTCOMES:
glucose metabolism | Before four months intervention.
  Glucose metabolism will be estimated by an oral glucose tolerance test (OGTT).
weight | Before intervention.
weight | after four months intervention.
glucose metabolism | Before intervention.
  Glucose metabolism will be estimated by an oral glucose tolerance test (OGTT).

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Ruige, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium